CLINICAL TRIAL: NCT03698357
Title: Effect of Interactive Video Balance-based Exercise in Persons With Stroke
Brief Title: Video Balance-based Exercise in Persons With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Lai chien hung, Professor, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201708024
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2018-10

CONDITIONS: Stroke
Keywords: interactive video balance-based exercise; conventional physiotherapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive video balance-based exercise (Experimental): Fifteen participants in group A will undergo 30 minutes a day and 3 days a week interactive video balance-based exercise intervention for four weeks.
  Interventions: Behavioral: interactive video balance-based exercise
- Conventional physiotherapy (Active Comparator): Another 15 participants allocated to the group B will receive 30 minutes a day and 3 days a week conventional rehabilitation for four weeks.
  Interventions: Behavioral: Conventional physiotherapy

INTERVENTIONS:
Behavioral: interactive video balance-based exercise — Interactive video balance-based exercise :10 minutes of warm up exercise, 30 minutes of Interactive video balance-based exercise and 5 minutes of cool down exercise.
  Arms: Interactive video balance-based exercise
Behavioral: Conventional physiotherapy — conventional physiotherapy: 10 minutes of warm up exercise, 30 minutes conventional physiotherapy and 5 minutes of cool down exercise. Conventional physiotherapy contains rolling, sitting, balance exercise, standing, overground walking, facilitation of the paretic limbs, and so on.
  Arms: Conventional physiotherapy

SUMMARY:
This study is to compare the effects of Interactive video balance-based exercise (IVBE) intervention and conventional rehabilitation on the balance and functional performance in stroke survivors. Fifteen participants will receive Interactive video balance-based exercise, while the other half will receive conventional rehabilitation.

DETAILED DESCRIPTION:
Thirty individuals with stroke are recruited and allocated to 2 groups in this study. Fifteen participants in group A will undergo 30 minutes a day and 3 days a week interactive video balance-based exercise intervention for four weeks. Another 15 participants allocated to the group B will receive 30 minutes a day and 3 days a week conventional rehabilitation for four weeks. Time up go test (TUG), Berg Balance Scale (BBS), Modified Falls Efficacy Scale (MFES), Motricity Index (MI), Functional Ambulation Category (FAC) were assessed before and after intervention in both groups

ELIGIBILITY:
Inclusion Criteria:

1. patients present with unilateral hemiplegia caused by a first-ever stroke
2. cognitive ability is sufficient to understand the nature of study (Mini-Mental State Examination score>=23)
3. medical and psychological condition stable

Exclusion Criteria:

1. patients having severe spasticity (Modified Ashworth scale > 3)
2. severe hearing or eye problem
3. intake of drugs or other medical condition that can affect function or can't tolerate rehabilitation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Change of Berg Balance Scale (BBS) | Measurement before and after intervention ( week 0 and at the end of week 4) in both groups
  Participants perform a series of 14 functional balance tasks, such as maintaining a quiet stance, sitting-to-stand, shifting weight and reaching, turning in place, standing on one leg, and maintaining a tandem stance.

SECONDARY OUTCOMES:
Change of Time Up Go test (TUG) | Measurement before and after intervention ( week 0 and at the end of week 4) in both groups
  The TUG test is a quick, reliable, valid, and accurate method commonly used to test dynamic stability and functional mobility. In the test, participants stand up from a 46-cm-high armchair with back support, walk straight for 3 m, turn around, walk back to the chair, and sit down as quickly and safely as possible.
Change of Modified Falls Efficacy Scale (MFES) | Measurement before and after intervention ( week 0 and at the end of week 4) in both groups
  The MFES is a 14-item rating scale questionnaire that contains the original 10-activity Falls Efficacy Scale and 4 additional activities. It is used to assess confidence of not falling while performing daily activities.
Change of Motricity Index (MI) | Measurement before and after intervention ( week 0 and at the end of week 4) in both groups
  The MI reflects general muscle strength in persons with stroke.
Change of Functional Ambulation Category (FAC) | Measurement before and after intervention ( week 0 and at the end of week 4) in both groups
  The FAC is based on the required level of assistance during walking in individuals with stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hung Lai, MD PhD, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical university Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen SC, Lin CH, Su SW, Chang YT, Lai CH. Feasibility and effect of interactive telerehabilitation on balance in individuals with chronic stroke: a pilot study. J Neuroeng Rehabil. 2021 Apr 26;18(1):71. doi: 10.1186/s12984-021-00866-8. PMID 33902646